CLINICAL TRIAL: NCT00754845
Title: A Double Blind Randomization to Letrozole or Placebo for Women Previously Diagnosed With Primary Breast Cancer Completing Five Years of Adjuvant Aromatase Inhibitor Either as Initial Therapy or After Tamoxifen (Including Those in The MA.17 Study)
Brief Title: Letrozole in Breast Cancer Who Have Received 5 Years of Aromatase Inhibitor Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network); Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA17R; CAN-NCIC-MA17R (Registry Identifier: NCI US - Physician Data Query); CDR0000614819 (Other: PDQ)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Experimental): Patients receive oral letrozole once daily for up to 5 years in the absence of unacceptable toxicity, disease recurrence, or development of a second malignancy.
  Interventions: Drug: letrozole
- Placebo (Placebo Comparator): Patients receive oral placebo once daily for up to 5 years in the absence of unacceptable toxicity, disease recurrence, or development of a second malignancy.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: letrozole — Given orally
  Other Names: femara
  Arms: Letrozole
Other: placebo — Given orally
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether letrozole is more effective than a placebo in treating in women with breast cancer who have already received 5 years of aromatase inhibitor therapy.

PURPOSE: This randomized phase III trial is studying letrozole to see how well it works compared with a placebo in treating women with primary breast cancer who have received 5 years of aromatase inhibitor therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the disease-free survival of women with primary breast cancer treated with letrozole vs placebo after completing approximately 5 years (i.e., 4½ - 6 years) of aromatase inhibitor therapy (e.g., letrozole, anastrozole, or exemestane).

Secondary

* To compare the effect of these drugs on overall (all cause specific) mortality of these patients.
* To compare the incidence of contralateral breast cancer in patients treated with these drugs.
* To evaluate the long-term clinical and laboratory safety of aromatase inhibitor therapy, particularly cardiovascular morbidity and mortality (e.g., significant coronary artery disease, including myocardial infarction and angina requiring percutaneous transluminal coronary angioplasty or coronary artery bypass graft, fatal and nonfatal strokes, and all vascular deaths); incidence of all bone fractures (with particular emphasis on hip and wrist fractures as indicators of osteoporosis); changes in bone density; and common toxicities.
* To compare overall quality of life (QOL) and menopausal-specific QOL of patients treated with these drugs.

OUTLINE: This is a multicenter study. Patients are stratified according to lymph node status at diagnosis (negative vs positive vs unknown), prior adjuvant chemotherapy (yes vs no), interval between last dose of aromatase inhibitor therapy and study randomization (< 6 months vs 6 months to 2 years), and duration of prior tamoxifen citrate use (0 vs < 2 years vs 2 - 4½ years vs > 4½ years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral letrozole once daily for up to 5 years in the absence of unacceptable toxicity, disease recurrence, or development of a second malignancy.
* Arm II: Patients receive oral placebo once daily for up to 5 years in the absence of unacceptable toxicity, disease recurrence, or development of a second malignancy.

Patients undergo bone mineral density measurement by DEXA scan at baseline (if not done within 12 months of study entry), at 24 and 48 months during study therapy, and at the completion of study therapy. Some patients also complete quality-of-life questionnaires at baseline and at 12, 24, 36, 48, and 60 months.

After completion of study therapy, patients are followed annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously diagnosed with primary breast cancer
* Must have received 4½ - 6 years of aromatase inhibitor therapy (e.g., letrozole, anastrozole, or exemestane), either as initial therapy or after prior tamoxifen citrate, including treatment received as part of clinical trial CAN-NCIC-MA17

  * Completed aromatase inhibitor therapy ≤ 2 years ago
* No metastatic or recurrent disease, contralateral breast cancer, or ductal carcinoma in situ in either breast, as determined by the following:

  * Clinical examination of the breast area, axillae, and neck within the past 60 days
  * Mammogram within the past 12 months*
  * Chest x-ray within the past 60 days
  * Bone scan, if alkaline phosphatase > 2 times normal and/or there are symptoms of metastatic disease AND confirmatory x-ray, if bone scan results are questionable, within the past 60 days
  * Abdominal ultrasound, liver scan, or CT scan of the abdomen within the past 60 days, if ALT, AST, or alkaline phosphatase > 2 times normal NOTE: *A baseline mammogram is not required for patients who have undergone bilateral complete mastectomy
* Hormone-receptor status:

  * Estrogen receptor positive (ER+) and/or progesterone receptor positive (PR+) primary tumor at the time of diagnosis, defined as a tumor receptor content of > 10 fmol/mg protein or receptor positive by immunocytochemical assay (for patients not previously enrolled on clinical trial CAN-NCIC-MA17)
  * ER+ and/or PR+ primary tumor OR hormone receptor status of primary tumor unknown (for patients previously enrolled on clinical trial CAN-NCIC-MA17)

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 5 years
* WBC > 3.0 x 10^9/L OR granulocyte count (polymorphs + bands) ≥ 1.5 times 10^9/L
* Platelet count > 100 x 10^9/L
* AST and/or ALT < 2 times upper limit of normal (ULN)*
* Alkaline phosphatase < 2 times ULN*
* Able (i.e. sufficiently fluent) and willing to complete quality-of-life questionnaires in either English or French (NCIC CTG participating centers)

  * Inability to complete questionnaires due to illiteracy in English or French, loss of sight, or other equivalent reason allowed
* Accessible for treatment and follow-up
* No other prior or concurrent malignancy except adequately treated, superficial squamous cell or basal cell skin cancer, carcinoma in situ of the cervix, or other cancer treated > 5 years ago that is presumed cured NOTE: *Elevated levels allowed provided imaging examinations have ruled out metastatic disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent selective estrogen receptor modulator (e.g., raloxifene, idoxifene)
* No other concurrent anticancer therapy

Ages: 0 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1918 (Actual)
Dates: Start 2004-11-23 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (43):
- Canada (42):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Centre de Sante et de services sociaux de Gatineau, Gatineau, Quebec
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - L'Hotel-Dieu de Levis, Lévis, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUM - Hotel Dieu du Montreal, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Wythenshawe Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goss PE, Ingle JN, Pritchard KI, Robert NJ, Muss H, Gralow J, Gelmon K, Whelan T, Strasser-Weippl K, Rubin S, Sturtz K, Wolff AC, Winer E, Hudis C, Stopeck A, Beck JT, Kaur JS, Whelan K, Tu D, Parulekar WR. Extending Aromatase-Inhibitor Adjuvant Therapy to 10 Years. N Engl J Med. 2016 Jul 21;375(3):209-19. doi: 10.1056/NEJMoa1604700. Epub 2016 Jun 5. PMID 27264120
- [Derived] Li Y, Zheng X, Tu D, Ingle JN, Goss PE, Parulekar WR, Qin G. Predicting the clinical outcomes and benefit from letrozole after 5 years of treatment with aromatase inhibitors for early breast cancer: analysis from CCTG MA.17R. Breast Cancer Res Treat. 2022 Feb;191(3):523-533. doi: 10.1007/s10549-021-06448-5. Epub 2021 Nov 26. PMID 34825307
- [Derived] Ethier JL, Anderson GM, Austin PC, Clemons M, Parulekar W, Shepherd L, Summers Trasiewicz L, Tu D, Amir E. Influence of the competing risk of death on estimates of disease recurrence in trials of adjuvant endocrine therapy for early-stage breast cancer: A secondary analysis of MA.27, MA.17 and MA.17R. Eur J Cancer. 2021 May;149:117-127. doi: 10.1016/j.ejca.2021.02.034. Epub 2021 Apr 11. PMID 33853037
- [Derived] Lemieux J, Brundage MD, Parulekar WR, Goss PE, Ingle JN, Pritchard KI, Celano P, Muss H, Gralow J, Strasser-Weippl K, Whelan K, Tu D, Whelan TJ. Quality of Life From Canadian Cancer Trials Group MA.17R: A Randomized Trial of Extending Adjuvant Letrozole to 10 Years. J Clin Oncol. 2018 Feb 20;36(6):563-571. doi: 10.1200/JCO.2017.75.7500. Epub 2018 Jan 12. PMID 29328860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Letrozole | Placebo
Started | 959 | 959
Completed | 959 | 959
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Placebo | Total
Number analyzed (Participants) | 959 | 959 | 1918
Age, Continuous [Median (Full Range); unit: years] | 65.6 [43 to 92.2] | 64.8 [43.4 to 89.9] | 65.1 [43 to 92.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 959 | 959 | 1918
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 940 | 939 | 1879
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 276 | 285 | 561
  United States | 683 | 674 | 1357
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    Grade 0 | 852 | 856 | 1708
    Grade 1 | 100 | 95 | 195
    Grade 2 | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: It is defined as the months from the day of randomization to the earliest date when a recurrence of the primary disease (recurrence in the breast, chest wall and nodal sites or the development of metastatic disease) or a contralateral breast cancer was observed. Subjects who died without recurrence of the primary disease or the development of the contralateral breast cancer were censored at their death date. If a patient has not recurred, developed a contralateral breast cancer, or died, disease-free survival was censored on the date of the last day the patient was known to be alive. Probability of disease free survival at 5 years is estimated and reported.
Time Frame: Unitil the end of study with a median follow up of 75 months
Population: All women randomized were included in the analysis based on treatment arm they were randomized.
Measure: Number (95% Confidence Interval); unit: probability of DFS at 5 years
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 959 | 959
probability of DFS at 5 years | 0.95 [0.93 to 0.96] | 0.91 [0.89 to 0.93]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.01, Log Rank; Stratified by the stratification factors at randomization; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.48 to 0.91]

2. Secondary Outcome: Incidence of Contralateral Breast Cancer
Description: The annual incidence rate was estimated based on the time to the development of contralateral breast cancer, which was calculated in months from the day of randomization to the diagnosis date of contralateral breast cancer for subjects who had developed the contralateral breast cancer, to the time of death for the patient who died, or to the last day the patient was known alive for subjects without contralateral breast cancer
Time Frame: 10 years
Population: All women randomized
Measure: Number (95% Confidence Interval); unit: Number of new case per 1000 person years
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 959 | 959
Number of new case per 1000 person years | 2.1 [1.0 to 3.2] | 4.9 [3.2 to 6.7]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.007, Log Rank

3. Secondary Outcome: Overall Survival (OS)
Description: For subjects who died, overall survival was calculated in months from the day of randomization to the date of death. Otherwise, survival was censored at the last day the patient was known to be alive. Probability of overall survival at 5 years is estimated and reported.
Time Frame: Until the end of study with a median follow-up of 75 months
Population: All women randomized
Measure: Number (95% Confidence Interval); unit: probability of OS at 5 years
Groups:
- Arm I: Patients receive oral letrozole once daily for up to 5 years in the absence of unacceptable toxicity, disease recurrence, or development of a second malignancy.
  letrozole: Given orally
- Arm II: Patients receive oral placebo once daily for up to 5 years in the absence of unacceptable toxicity, disease recurrence, or development of a second malignancy.
  placebo: Given orally
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 959 | 959
probability of OS at 5 years | 0.93 [0.92 to 0.95] | 0.94 [0.92 to 0.95]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.83, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.73 to 1.28]

4. Secondary Outcome: Change From Baseline in Role Function- Physical Scale on SF(Short Form)-36 Health Survey
Description: Difference between post baseline scores and baseline score of role function-physical scale on SF-36 Health Survey (scale range between 0 and 100 with higher score indicating better quality of life).
Time Frame: 8 years
Population: All randomized patients.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 959 | 959
score on a scale | -7.74 (1.09) | -6.28 (1.08)
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p < 0.01, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: During protocol treatment of 5 years
Arm/Group | Arm I | Arm II
All-Cause Mortality (participants affected / at risk) | 100/959 | 100/954
Serious Adverse Events (participants affected / at risk) | 15/959 | 19/954
Other Adverse Events (participants affected / at risk) | 863/959 | 841/954
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=959) | Arm II (N=954)
Cardiac troponin I (cTnI) (Cardiac disorders) | 0 | 1
Thrombosis/embolism (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Constitutional Symptoms - Other (General disorders) | 0 | 1
Creatinine (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 2
CNS hemorrhage/bleeding (Blood and lymphatic system disorders) | 0 | 1
Melena/GI bleeding (Blood and lymphatic system disorders) | 1 | 0
Rectal bleeding/ hematochezia (Blood and lymphatic system disorders) | 1 | 0
Liver dysfunction/ failure (clinical) (Hepatobiliary disorders) | 1 | 0
Hepatic - Other (Hepatobiliary disorders) | 1 | 0
Infection without neutropenia (Infections and infestations) | 2 | 3
Infection with unknown ANC (Infections and infestations) | 0 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 3
Neuropathy-motor (Nervous system disorders) | 0 | 1
Sudden death (General disorders) | 4 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Second malignacy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ ventricular tachycardia) (Cardiac disorders) | 1 | 1
Edema (Cardiac disorders) | 1 | 0
Cardiac left ventricular function (Cardiac disorders) | 1 | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 4
Supraventricular arrhythmias (SVT/atrial fibrillation/ flutter) (Cardiac disorders) | 1 | 0
Cardiovascular/ General - Other (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=959) | Arm II (N=954)
Edema (Cardiac disorders) | 158 | 136
Hypertension (Cardiac disorders) | 157 | 145
Hot flashes/ flushes (Endocrine disorders) | 360 | 354
Fatigue (General disorders) | 346 | 355
Sweating (General disorders) | 176 | 175
Anorexia (Gastrointestinal disorders) | 46 | 52
Constipation (Gastrointestinal disorders) | 117 | 140
Diarrhea (Gastrointestinal disorders) | 105 | 81
Dyspepsia/heartburn (Gastrointestinal disorders) | 86 | 79
Nausea (Gastrointestinal disorders) | 69 | 76
Infection w/o neutropenia (Infections and infestations) | 81 | 82
Arthritis (Musculoskeletal and connective tissue disorders) | 317 | 288
Hypercholesterolemia (Metabolism and nutrition disorders) | 203 | 184
Hyperglycemia (Metabolism and nutrition disorders) | 56 | 66
Anxiety (Nervous system disorders) | 54 | 56
Dizziness (Nervous system disorders) | 145 | 139
Insomnia (Nervous system disorders) | 269 | 243
Depression (Nervous system disorders) | 152 | 150
Neuropathy-sensory (Nervous system disorders) | 110 | 107
Abdominal pain (General disorders) | 51 | 38
Headache (General disorders) | 151 | 138
Arthralgia (General disorders) | 513 | 475
Myalgia (General disorders) | 268 | 240
Bone pain (General disorders) | 174 | 133
Pain-Other (General disorders) | 73 | 77
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 69
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 148 | 165
Alopecia (Skin and subcutaneous tissue disorders) | 61 | 64
Vaginal dryness (Reproductive system and breast disorders) | 102 | 96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No